CLINICAL TRIAL: NCT02968914
Title: A Multicenter, Randomized, Open-Label, Parallel Group Phase 1 Pharmacokinetic Comparability Study of Benralizumab Administrated Using Accessorized Pre-Filled Syringe (APFS) or Autoinjector (AI) in Healthy Volunteers.
Brief Title: Pharmacokinetic Comparability of Benralizumab Using Accessorized Pre-Filled Syringe or Autoinjector in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D3250C00030
Record Dates: First submitted 2016-10-28; First posted 2016-11-21 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-06

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease
Keywords: Asthma; Chronic Obstructive pulmonary Disease; Pharmacokinetics; Healthy volunteers
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive | interventions — benralizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Benralizumab by Accessorized Pre-Filled Syringe (Active Comparator): Drug administration by Accessorized Pre-Filled Syringe. A total of 180 subjects will be randomized and will be stratified by weight group (55 to 69.9 kg, 70 to 84.9 kg and 85 to 100 kg). Within each of the 3 weight groups, subjects will be randomized 1:1:1:1:1:1 to 1 of the 6 combinations of treatment (APFS) with injection site (upper arm, abdomen or thigh)
  Interventions: Biological: Benralizumab
- Benralizumab by Autoinjector (Other): Drug administration by Autoinjector A total of 180 subjects will be randomized and will be stratified by weight group (55 to 69.9 kg, 70 to 84.9 kg and 85 to 100 kg). Within each of the 3 weight groups, subjects will be randomized 1:1:1:1:1:1 to 1 of the 6 combinations of treatment (APFS) with injection site (upper arm, abdomen or thigh)
  Interventions: Biological: Benralizumab

INTERVENTIONS:
Biological: Benralizumab — A humanized, afucosylated, monoclonal antibody (mAb) that binds specifically to the human IL-5 receptor alpha subunit (IL-5Rα) on the target cell.
  Arms: Benralizumab by Accessorized Pre-Filled Syringe
Biological: Benralizumab — A humanized, afucosylated, monoclonal antibody (mAb) that binds specifically to the human IL-5 receptor alpha subunit (IL-5Rα) on the target cell.
  Arms: Benralizumab by Autoinjector

SUMMARY:
An open-label, single dose Pharmacokinetic (PK) comparability study to demonstrate comparable drug exposure following Subcutaneous benralizumab administration by using accessorized pre-filled syringe (APFS) or autoinjector (AI) devices.

DETAILED DESCRIPTION:
A study of descriptive comparison of benralizumab PK by weight and injection site.

This study will be a multicenter, randomized, open-label, parallel group Phase 1 study designed to compare benralizumab PK exposure in healthy subjects following single subcutaneous (SC) administration of fixed 30 mg dose of benralizumab by using APFS and single-use AI. Eligible subjects will be healthy subjects aged 18 to 55 years, with a body weight of 55 to 100 kg and a body mass index of 18 to 29.9 kg/m2 . A total of 180 subjects will be randomized. Randomization will be stratified by weight group (55 to 69.9 kg, 70 to 84.9 kg and 85 to 100 kg), and within each of the 3 weight groups, subjects will be randomized 1:1:1:1:1:1 to 1 of the 6 combinations of treatment (APFS or AI) with injection site (upper arm, abdomen or thigh), presented in Table 1. This study will be performed at 2 study centers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non-child-bearing potential aged 18 to 55 years (inclusive) with suitable veins for cannulation or repeated venipuncture.
* Females must be non pregnant,non lactating and non-child-bearing potential, confirmed at screening
* Sexually active male willingness to use contraception
* Body mass index (BMI) between 18 and 29.9 kg/m2 inclusive and weigh at least 55 kg and no more than 100 kg inclusive.

Exclusion Criteria:

* History of any clinically significant disease, severe allergy/anaphylaxis to any biologic therapy, Guillain-Barré syndrome, smoking and alcohol or drug abuse
* Diagnosis of helminth parasitic infection and acute upper or lower respiratory infections
* Disorders related to cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, hematological, psychiatric, or major physical impairment
* Alanine aminotransferase/aspartate aminotransferase level ≥1.5 times the upper limit of normal
* White blood cell count and neutrophils < lower limit of normal
* Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of Investigational medicinal product (IMP)
* Positive result for serum hepatitis B surface antigen or anti-Hemoglobin C (anti-HBc) antibody, hepatitis C antibody, and human immunodeficiency virus (HIV) antibody.
* Intake of new chemical entity (not been approved for marketing) within 3 months of the first administration of investigational product
* Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to screening
* Receipt of immunoglobulin or blood products within 30 days prior to the date informed consent
* Receipt of any marketed (e.g., omalizumab, mepolizumab etc.) or investigational biologic within 4 months or 5 half-lives prior to the date informed consent
* Receipt of live attenuated vaccines 30 days prior to randomization on Day 1
* Current malignancy, or history of malignancy except (basal cell carcinoma, localized squamous cell carcinoma of the skin or in situ carcinoma of the cervix)
* Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.
* Use of antacids, analgesics (except paracetamol/acetaminophen), herbal remedies, mega-dose vitamins (20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of IMP or longer
* Previous receipt of received benralizumab
* Any ongoing or recent minor medical complaints
* Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2017-07-13 (Actual); Study Completion 2017-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Rainard Fuhr, Medicine, Principal Investigator — PAREXEL Early Phase Clinical Unit Berlin; Dr. Pablo Forte-Soto, Principal Investigator — PAREXEL Early Phase Clinical Unit London
Locations (2):
- Germany (2):
  - Research Site, Berlin
  - Research Site, Harrow

REFERENCES:
- [Derived] Martin UJ, Fuhr R, Forte P, Barker P, Axley MJ, Aurivillius M, Yan L, Roskos L. Comparison of autoinjector with accessorized prefilled syringe for benralizumab pharmacokinetic exposure: AMES trial results. J Asthma. 2021 Jan;58(1):93-101. doi: 10.1080/02770903.2019.1663428. Epub 2019 Sep 20. PMID 31539289
- See also: SAP — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4091&filename=230172_D3250C00030_SAP_Final_21-Sep-2018.pdf
- See also: SP — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4091&filename=230172_D3250C00030_Protocol_Final_21-Sep-2018.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who met all the inclusion and none of the exclusion criteria were enrolled at PAREXEL Early Phase Clinical Unit in Berlin and London.
Pre-assignment Details: Subjects attended a Screening Visit within 28 days before receiving their first dose of Benralizumab. All subjects underwent inclusion exclusion criteria assessment and all eligible subjects signed the informed consent before undergoing any study-related procedures.
Groups:
- Benralizumab 30mg Autoinjector (AI): All randomized subjects received 30mg Benralizumab by AI under fasted conditions.
- Benralizumab 30mg Accessorized Pre-filled Syringe (AFPS): All randomized subjects received 30mg Benralizumab by APFS under fasted conditions.
Period: Overall Study
Arm/Group | Benralizumab 30mg Autoinjector (AI) | Benralizumab 30mg Accessorized Pre-filled Syringe (AFPS)
Started | 90 | 90
Completed | 90 | 90
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Benralizumab 30mg Autoinjector (AI) | Benralizumab 30mg Accessorized Pre-filled Syringe (AFPS) | Total
Number analyzed (Participants) | 90 | 90 | 180
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.8 (10.8) | 41.1 (11.1) | 40.9 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 33
  Male | 73 | 74 | 147
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 89 | 88 | 177
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 5 | 10
  White | 83 | 80 | 163
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From Zero to Infinity (AUCinf)
Description: To compare the AUCinf following single SC administration of Benralizumab by using APFS or AI devices
Time Frame: At Pre-dose (Day 1) and at Days 2, 4, 5, 6, 8, 15, 29, 43 and 57
Population: The PK analysis set consisted of all subjects who received benralizumab for whom PK blood samples were assumed not to be affected by factors such as protocol violations (e.g., disallowed medications or incomplete dose administration) and who had at least one post dose quantifiable serum PK observation.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day·ng/mL
Groups:
- Benralizumab 30mg AI: All randomized subjects received 30mg Benralizumab by AI under fasted conditions.
- Benralizumab 30mg AFPS: All randomized subjects received 30mg Benralizumab by APFS under fasted conditions.
Arm/Group | Benralizumab 30mg AI | Benralizumab 30mg AFPS
Number analyzed (Participants) | 88 | 87
day·ng/mL | 72210 (29.7) | 76220 (32.1)
Statistical Analysis 1: Comparison: Benralizumab 30mg AI vs Benralizumab 30mg AFPS; Test type: Superiority; ANOVA; Geometric mean ratio (%) = 94.46, 90% CI 2-sided [88.16 to 101.21]

2. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to Time of Last Quantifiable Concentration (AUClast)
Description: To compare the AUClast following single SC administration of Benralizumab by using APFS or AI devices
Time Frame: At Pre-dose (Day 1) and at Days 2, 4, 5, 6, 8, 15, 29, 43 and 57
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day·ng/mL
Arm/Group | Benralizumab 30mg AI | Benralizumab 30mg AFPS
Number analyzed (Participants) | 90 | 90
day·ng/mL | 60560 (27.3) | 65230 (29.2)
Statistical Analysis 1: Comparison: Benralizumab 30mg AI vs Benralizumab 30mg AFPS; Test type: Superiority; ANOVA; Geometric mean ratio (%) = 92.83, 90% CI 2-sided [87.41 to 98.58]

3. Primary Outcome: Maximum Observed Concentration (Cmax)
Description: To compare the Cmax following single SC administration of Benralizumab by using APFS or AI devices
Time Frame: At Pre-dose (Day 1) and at Days 2, 4, 5, 6, 8, 15, 29, 43 and 57
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Benralizumab 30mg AI | Benralizumab 30mg AFPS
Number analyzed (Participants) | 90 | 90
ng/mL | 2096 (32.7) | 2269 (35.4)
Statistical Analysis 1: Comparison: Benralizumab 30mg AI vs Benralizumab 30mg AFPS; Test type: Superiority; ANOVA; Geometric mean ratio (%) = 92.34, 90% CI 2-sided [86.34 to 98.75]

4. Secondary Outcome: Time When Maximum Concentration is Observed (Tmax)
Description: To evaluate the Tmax of Benralizumab administered to various injection sites and in subjects with different body weight ranges
Time Frame: At Pre-dose (Day 1) and at Days 2, 4, 5, 6, 8, 15, 29, 43 and 57
Population: as for outcome 1
Measure: Median (Full Range); unit: Days
Arm/Group | Benralizumab 30mg AI | Benralizumab 30mg AFPS
Number analyzed (Participants) | 90 | 90
Days
  Abdomen 55.0 to 69.9 kg: number analyzed (Participants) | 10 | 10
  Abdomen 55.0 to 69.9 kg | 4.59 [2.97 to 7.04] | 6.06 [4.00 to 14.00]
  Abdomen 70.0 to 84.9 kg: number analyzed (Participants) | 10 | 10
  Abdomen 70.0 to 84.9 kg | 6.98 [3.98 to 14.00] | 5.98 [2.95 to 14.05]
  Abdomen 85.0 to 100.0 kg: number analyzed (Participants) | 10 | 10
  Abdomen 85.0 to 100.0 kg | 5.06 [3.95 to 7.11] | 6.96 [3.99 to 7.10]
  Thigh 55.0 to 69.9 kg: number analyzed (Participants) | 10 | 10
  Thigh 55.0 to 69.9 kg | 4.00 [2.97 to 7.01] | 4.52 [2.94 to 7.04]
  Thigh 70.0 to 84.9 kg: number analyzed (Participants) | 10 | 10
  Thigh 70.0 to 84.9 kg | 4.05 [2.98 to 6.90] | 3.52 [2.95 to 7.12]
  Thigh 85.0 to 100.0 kg: number analyzed (Participants) | 10 | 10
  Thigh 85.0 to 100.0 kg | 4.59 [2.94 to 13.95] | 4.03 [2.98 to 6.98]
  Upper arm 55.0 to 69.9 kg: number analyzed (Participants) | 10 | 10
  Upper arm 55.0 to 69.9 kg | 6.97 [3.97 to 14.02] | 4.96 [3.02 to 14.04]
  Upper arm 70.0 to 84.9 kg: number analyzed (Participants) | 10 | 10
  Upper arm 70.0 to 84.9 kg | 7.00 [5.01 to 14.03] | 5.02 [2.99 to 8.01]
  Upper arm 85.0 to 100.0 kg: number analyzed (Participants) | 10 | 10
  Upper arm 85.0 to 100.0 kg | 7.00 [3.09 to 14.03] | 6.97 [1.02 to 14.13]

5. Secondary Outcome: Terminal Half-life (t½)
Description: To evaluate the t½ of Benralizumab administered to various anatomical injection sites and in subjects with different body weight ranges.
Time Frame: At Pre-dose (Day 1) and at Days 2, 4, 5, 6, 8, 15, 29, 43 and 57
Population: The PK analysis set consisted of all the subjects as defined for above endpoint. For Benralizumab 30mg AI, two subjects and for Benralizumab 30mg AFPS, three subjects were excluded from the PK analysis set.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days
Arm/Group | Benralizumab 30mg AI | Benralizumab 30mg AFPS
Number analyzed (Participants) | 88 | 87
Days
  Abdomen 55.0 to 69.9 kg: number analyzed (Participants) | 10 | 9
  Abdomen 55.0 to 69.9 kg | 18.83 (24.9) | 20.15 (21.8)
  Abdomen 70.0 to 84.9 kg: number analyzed (Participants) | 10 | 10
  Abdomen 70.0 to 84.9 kg | 20.22 (21.0) | 17.43 (21.7)
  Abdomen 85.0 to 100.0 kg: number analyzed (Participants) | 10 | 10
  Abdomen 85.0 to 100.0 kg | 19.59 (19.9) | 21.04 (21.7)
  Thigh 55.0 to 69.9 kg: number analyzed (Participants) | 10 | 10
  Thigh 55.0 to 69.9 kg | 18.58 (20.6) | 19.72 (21.4)
  Thigh 70.0 to 84.9 kg: number analyzed (Participants) | 10 | 10
  Thigh 70.0 to 84.9 kg | 19.93 (23.4) | 18.28 (17.9)
  Thigh 85.0 to 100.0 kg: number analyzed (Participants) | 9 | 10
  Thigh 85.0 to 100.0 kg | 19.02 (19.9) | 17.30 (11.5)
  Upper arm 55.0 to 69.9 kg: number analyzed (Participants) | 10 | 8
  Upper arm 55.0 to 69.9 kg | 22.46 (13.6) | 17.30 (26.9)
  Upper arm 70.0 to 84.9 kg: number analyzed (Participants) | 10 | 10
  Upper arm 70.0 to 84.9 kg | 20.54 (14.0) | 20.16 (25.3)
  Upper arm 85.0 to 100.0 kg: number analyzed (Participants) | 9 | 10
  Upper arm 85.0 to 100.0 kg | 19.01 (26.9) | 19.42 (26.3)

6. Secondary Outcome: Apparent Extravascular Clearance (CL/F)
Description: To evaluate the CL/F of Benralizumab administered to various anatomical injection sites and in subjects with different body weight ranges.
Time Frame: At Pre-dose (Day 1) and at Days 2, 4, 5, 6, 8, 15, 29, 43 and 57
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/day
Arm/Group | Benralizumab 30mg AI | Benralizumab 30mg AFPS
Number analyzed (Participants) | 88 | 87
mL/day
  Abdomen 55.0 to 69.9 kg: number analyzed (Participants) | 10 | 9
  Abdomen 55.0 to 69.9 kg | 388.8 (34.3) | 388.9 (43.8)
  Abdomen 70.0 to 84.9 kg: number analyzed (Participants) | 10 | 10
  Abdomen 70.0 to 84.9 kg | 462.9 (29.5) | 508.9 (33.2)
  Abdomen 85.0 to 100.0 kg: number analyzed (Participants) | 10 | 10
  Abdomen 85.0 to 100.0 kg | 504.6 (18.3) | 402.7 (30.4)
  Thigh 55.0 to 69.9 kg: number analyzed (Participants) | 10 | 10
  Thigh 55.0 to 69.9 kg | 350.1 (32.6) | 281.1 (16.8)
  Thigh 70.0 to 84.9 kg: number analyzed (Participants) | 10 | 10
  Thigh 70.0 to 84.9 kg | 393.7 (29.6) | 325.9 (18.2)
  Thigh 85.0 to 100.0 kg: number analyzed (Participants) | 9 | 10
  Thigh 85.0 to 100.0 kg | 378.2 (26.8) | 406.0 (22.9)
  Upper arm 55.0 to 69.9 kg: number analyzed (Participants) | 10 | 8
  Upper arm 55.0 to 69.9 kg | 345.8 (24.7) | 455.2 (29.8)
  Upper arm 70.0 to 84.9 kg: number analyzed (Participants) | 10 | 10
  Upper arm 70.0 to 84.9 kg | 429.4 (19.5) | 366.1 (27.0)
  Upper arm 85.0 to 100.0 kg: number analyzed (Participants) | 9 | 10
  Upper arm 85.0 to 100.0 kg | 532.6 (21.7) | 471.6 (20.3)

7. Secondary Outcome: Apparent Volume of Distribution Based on the Terminal Phase (Vz/F)
Description: To evaluate the Vz/F of Benralizumab administered to various anatomical injection sites and in subjects with different body weight ranges.
Time Frame: At Pre-dose (Day 1) and at Days 2, 4, 5, 6, 8, 15, 29, 43 and 57
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Benralizumab 30mg AI | Benralizumab 30mg AFPS
Number analyzed (Participants) | 88 | 87
Liters
  Abdomen 55.0 to 69.9 kg: number analyzed (Participants) | 10 | 9
  Abdomen 55.0 to 69.9 kg | 10.56 (28.0) | 11.30 (28.4)
  Abdomen 70.0 to 84.9 kg: number analyzed (Participants) | 10 | 10
  Abdomen 70.0 to 84.9 kg | 13.50 (30.4) | 12.79 (25.5)
  Abdomen 85.0 to 100.0 kg: number analyzed (Participants) | 10 | 10
  Abdomen 85.0 to 100.0 kg | 14.26 (25.0) | 12.22 (15.8)
  Thigh 55.0 to 69.9 kg: number analyzed (Participants) | 10 | 10
  Thigh 55.0 to 69.9 kg | 9.386 (18.2) | 7.999 (15.5)
  Thigh 70.0 to 84.9 kg: number analyzed (Participants) | 10 | 10
  Thigh 70.0 to 84.9 kg | 11.32 (23.5) | 8.596 (13.5)
  Thigh 85.0 to 100.0 kg: number analyzed (Participants) | 9 | 10
  Thigh 85.0 to 100.0 kg | 10.38 (20.2) | 10.13 (21.0)
  Upper arm 55.0 to 69.9 kg: number analyzed (Participants) | 10 | 8
  Upper arm 55.0 to 69.9 kg | 11.21 (21.2) | 11.36 (17.7)
  Upper arm 70.0 to 84.9 kg: number analyzed (Participants) | 10 | 10
  Upper arm 70.0 to 84.9 kg | 12.72 (23.6) | 10.65 (18.7)
  Upper arm 85.0 to 100.0 kg: number analyzed (Participants) | 9 | 10
  Upper arm 85.0 to 100.0 kg | 14.61 (23.0) | 13.21 (32.9)

8. Secondary Outcome: Number of Participants With Adverse Events
Description: To evaluate safety and tolerability of Benralizumab
Time Frame: At predose and 2 h postdose (Day 1), Days 2, 4, 5, 6, 8, 15, 29, 43 and 57
Population: Safety set consisted of all subjects who received at least 1 dose of Benralizumab were included in the safety analysis for the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab 30mg AI | Benralizumab 30mg AFPS
Number analyzed (Participants) | 90 | 90
Participants
  Any AE | 50 | 46
  Death | 0 | 0
  Any SAE | 0 | 0
  Any AE leading to discontinuation | 0 | 0

9. Secondary Outcome: Antidrug Antibody (ADA) Status
Description: To evaluate the immunogenicity of Benralizumab
Time Frame: At predose (Day 1), Days 29 and 57
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab 30mg AI | Benralizumab 30mg AFPS
Number analyzed (Participants) | 90 | 90
Participants
  ADA prevalence (positive at any visit) | 2 | 6
  ADA incidence | 0 | 3

ADVERSE EVENTS:
Time Frame: At pre-dose and 2 h post-dose (Day 1), Days 2, 4, 5, 6, 8, 15, 29, 43 and 57
Arm/Group | Benralizumab 30mg Autoinjector (AI) | Benralizumab 30mg Accessorized Pre-filled Syringe (AFPS)
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/90
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/90
Other Adverse Events (participants affected / at risk) | 50/90 | 46/90
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Benralizumab 30mg Autoinjector (AI) (N=90) | Benralizumab 30mg Accessorized Pre-filled Syringe (AFPS) (N=90)
Nasopharyngitis (Infections and infestations) | 18 | 13
Rhinitis (Infections and infestations) | 2 | 0
Gingivitis (Infections and infestations) | 1 | 0
Myringitis (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Headache (Nervous system disorders) | 14 | 5
Dizziness (Nervous system disorders) | 2 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1
Hypertonia (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Tension headache (Nervous system disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 4 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Fatigue (General disorders) | 5 | 1
Influenza like illness (General disorders) | 1 | 1
Asthenia (General disorders) | 0 | 1
Discomfort (General disorders) | 0 | 1
Feeling hot (General disorders) | 1 | 0
Injection site hypersensitivity (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 2 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0
Haematoma (Vascular disorders) | 2 | 2
Insomnia (Psychiatric disorders) | 0 | 1
Listless (Psychiatric disorders) | 1 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Excessive cerumen production (Ear and labyrinth disorders) | 0 | 1
Eye pruritus (Eye disorders) | 1 | 0
Eye swelling (Eye disorders) | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 1
Cardiovascular symptom (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 1
Body temperature increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All clinical study findings and documents will be regarded as confidential. The investigator and members of his/her research team must not disclose such information without prior written approval from the sponsor.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-08-04): https://cdn.clinicaltrials.gov/large-docs/14/NCT02968914/SAP_000.pdf
  • Study Protocol (2017-07-07): https://cdn.clinicaltrials.gov/large-docs/14/NCT02968914/Prot_001.pdf